### **INFORMED CONSENT FORM**

Title: Multimodal Biomarker Predictors of Relapse in Major Depressive Disorder: A Hybrid

Retrospective-Prospective Cohort Study

NCT Number: Not yet available

**Document Date:** 01.12.2025

## **Prof. Dr. Mehmet Kemal Arıkan Psychiatry Clinic Informed Consent for Research Participation**

# When Should We Discontinue Antidepressant Treatment in Depression? A Prospective Observational Study

#### **Purpose and Method of the Study**

The data obtained from this study will form the basis for several future scientific investigations. If you agree to participate, you will undergo a series of electrophysiological assessments, clinical tests, and genetic analyses, which will require a blood sample. These evaluations may be repeated if clinically necessary.

These procedures do not pose any expected side effects. When you have recovered, your antidepressant treatment will be discontinued in accordance with the study protocol.

You will **not be charged any fees** for any procedure or follow-up related to this study.

### What are the benefits of participating?

The main benefit of this study is that the biological and electrophysiological measurements performed throughout the study will provide **clear and objective information** about your depression.

These results may help determine the most appropriate time to safely discontinue your medication.

#### What are the possible risks?

The most relevant risk is the possibility of experiencing withdrawal symptoms (such as dizziness, sleep disturbances, or fatigue) when your medication is discontinued as part of the study protocol. However, these symptoms are general and dissolve within a few weeks.

If you do not respond well or if any clinical deterioration occurs during discontinuation period, your previous treatment will be resumed immediately, and your participation in the study will be terminated.

#### Rights and Responsibilities of the Volunteer

- 1. Your participation in this research is entirely voluntary. You may refuse to take part or withdraw at any time without losing any rights and without facing any penalty or negative consequences.
- 2. All records that could reveal your identity will be kept strictly confidential and will not be disclosed publicly. Even if study results are published, your identity will remain anonymous.
- 3. Authorized national and international monitors, auditors, ethics committees, institutional officials, and relevant health authorities may access your original medical records when necessary. However, all data will remain confidential. By signing this consent form, you (or your legal representative) provide permission for such access.
- 4. If new information arises during the study that may affect your willingness to continue, you (or your legal representative) will be informed in a timely manner.
- 5. If you require further information about your rights or experience any adverse event related to the study, you may contact the individuals listed below 24 hours a day.

#### Consent

I have read and understood all the information provided in this Informed Consent Form. I have received written and verbal explanations regarding the study described above from the physician named below.

I voluntarily agree to participate in this research study and understand that I may withdraw from the study at any time, with or without providing a reason, and without any consequences.

I confirm that I am participating freely, without any pressure or coercion.

| Participant |
|----------------------|
| Name-Surname: |
| Date: |
| Signature: |
| Contact Information: |